CLINICAL TRIAL: NCT01129219
Title: Observation and Progressive Strength Training After Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Diakonhjemmet Hospital (Other)
Responsible Party: Mette Martinsen, Diakonhjemmet Sykehus
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1.2007.347
Record Dates: First submitted 2010-05-18; First posted 2010-05-24 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2007-03

CONDITIONS: Exercise
Keywords: Strength; Function; Mobility
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Usual care (Experimental): Subjects in the control group were asked to maintain their current lifestyle. No restrictions were placed on their exercise activities.
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Strength training — Strength training for 24 weeks

SUMMARY:
This is a randomized, controlled; single-blind parallel group trial carried out with hip fracture patients, starting at 12 weeks post fracture. Patients were approached during their acute stay in hospital, followed without any extra intervention for 12 weeks, and then randomized in a 2:1 manner to either intervention or control for the next 12 weeks. After the first 12 weeks intervention the intervention group were divided into two groups and randomized to an new single-blind parallel group trial for further intervention.

ELIGIBILITY:
Inclusion Criteria:at 12 weeks postoperative:

1. age at least 65 years
2. not living in nursing home
3. were able to undergo physical therapy for the hip fracture
4. scoring of 23 or more (out of 30) on the Mini Mental State Examination

Exclusion Criteria:

1. permanently institutionalized
2. had metastatic cancer
3. suffered from multi-trauma.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Bergs Balance scale | 24 weeks
  Bergs Balance Scale: The Berg balance scale (BBS) measures "functional balance," which has three dimensions: maintenance of a position, postural adjustment to voluntary movements, and reaction to external disturbance, scored 0-56 (Berg K. 1995).

SECONDARY OUTCOMES:
Strength | 24 weeks
  Secondary outcomes was the results on the Sit to Stand-test,which measure strength of lower limbs.

REFERENCES:
- [Result] Helen H Host, David R Sinacore, Kathryn L Bohnert, Karen Steger-May, Marybeth Brown and Ellen F Binder. Training-Induced Strength and Functional Adaptations After Hip Fracture. PHYS THER Vol. 87, No. 3, March 2007, pp. 292-303 Ellen F. Binder, MD; Marybeth Brown, PT, PhD; David R. Sinacore, PT, PhD; Karen Steger-May, MA; Kevin E. Yarasheski, PhD; Kenneth B. Schechtman. Effects of Extended Outpatient Rehabilitation After Hip Fracture. A Randomized Controlled Trial JAMA. 2004;292:837-846. Kathleen K Mangione, Rebecca L Craik, Susan S Tomlinson and Kerstin M Palombaro. Can Elderly Patients Who Have Had a Hip Fracture Perform Moderate- to High-Intensity Exercise at Home? PHYS THER Vol. 85, No. 8, August 2005, pp. 727-739 Klaus Hauer, Norbert Specht, Matthias Schuler, Peter Bärtsch1 and Peter Oster. Intensive physical training in geriatric patients after severe falls and hip surgery. Age and Ageing 2002; 31: 49-57 2002. David Moher1 , Kenneth F Schulz2 and Douglas G Altman. The CONSORT statement: revised recommendations for improving the quality of reports of parallel group randomized trials. BMC Medical Research Methodology 2001, 1:2doi:10.1186/1471-2288-1-2 Berg K, Wood-Dauphinee S, Williams JI. The Balance Scale: reliability assessment with elderly residents and patients with an acute stroke. Scand J Rehabil Med. 1995 Mar;27(1):27-36. Bohannon RW. Sit-to-stand test for measuring performance of lower extremity muscles. Percept Mot Skills. 1995 Feb;80(1):163-6. Podsiadlo D, Richardson S. The timed
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134